CLINICAL TRIAL: NCT05863390
Title: Effectiveness of McKenzie Exercises and Trochanteric Belt With Conventional Physical Therapy to Reduce Pain and Dysfunction of SI Joint in Pregnant Women
Brief Title: Effectiveness of McKenzie and Trochanteric Belt With CT Therapy to Reduce Pain and Dysfunction of SI Joint
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, DEAN, Superior University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall18/524
Record Dates: First submitted 2023-03-18; First posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Sacroiliac Joint Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- McKenzie exercise (Experimental)
  Interventions: Behavioral: McKenzie exercise
- Trochanteric belt (Other)
  Interventions: Diagnostic Test: Trochanteric belt

INTERVENTIONS:
Behavioral: McKenzie exercise — routine simple McKenzie exercise
  Arms: McKenzie exercise
Diagnostic Test: Trochanteric belt — Trochanteric belt with conventional physical therapy
  Arms: Trochanteric belt

SUMMARY:
To determine the effectiveness of McKenzie exercises and trochanteric belt with conventional physical therapy to reduce pain and dysfunction of Sacroiliac joint (SIJ) in pregnant women

DETAILED DESCRIPTION:
to findout the effectiveness of exercises in pregnant women

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients with sacroiliac joint pain are included and participant patients with age group 18- to 35
* low back pain due to sacroiliac joint who suffer from sever pain during sitting and during positioning change when stand from sitting position are included

Exclusion Criteria:

* Patients with age group of below 18 years and above 35 years
* Patients with disease of coagulopathy
* systemic infection
* skin infection over sacroiliac joint patients with history of allergies to injected medications.
* Patients with psoriasis
* inflammatory bowel disease
* peripheral arthritis
* Women with UTI complications are excluded.
* Women with respiratory issues are also excluded

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
feature of Visual analogue scale to check pain and feature PSFS to check Movement of joints | 6 Months
  Pre and Post interventions using VAS, PDFS

CONTACTS AND LOCATIONS:
Overall Officials: Abdul Wahab, Study Chair — Superior Uni
Locations (1):
- • General Hospital. • Chaudhary Muhammad Akram Teaching and Research Hospital, University of Lahore Teaching Hospital, Shadman Medical Center, Services Hospital, Bahria International Hospital, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No